CLINICAL TRIAL: NCT01176409
Title: VALacyclovir for Inflammation AttenuatioN Trial Pilot (VALIANT Pilot)
Brief Title: Can Valacyclovir Attenuate Inflammation in Antiretroviral-Treated HIV-Infected Individuals With Herpes Simplex Virus Type 2?
Acronym: VALIANT Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VALIANT-001
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Human Immunodeficiency Virus; Herpes Simplex
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose valacyclovir (Experimental): Valacyclovir 1g po BID
  Interventions: Drug: Valacyclovir
- Low dose valacyclovir (Active Comparator): Valacyclovir 500mg po BID
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator): Inert placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir will be used at two different dosages (1g po BID and 500mg po BID) to be used for 12 weeks. Supplied as 500mg caplets.
  Other Names: Apo-Valacycyclovir; Valtrex
  Arms: High dose valacyclovir; Low dose valacyclovir
Drug: Placebo — Placebo, supplied as caplets identical in appearance, odour and taste to valacyclovir 500mg caplets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the levels of immune and inflammatory markers among HIV-1, HSV-2 co-infected adults achieving plasma HIV RNA suppression to <50 copies/mL, between those randomized to valacyclovir and placebo, over a twelve-week intervention period.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has dramatically reduced HIV-1 infection (herein referred to as 'HIV') related morbidity and mortality, transforming an invariably fatal disease into a manageable, chronic condition. Yet even HAART-treated HIV infection is characterized by chronic systemic inflammation and immune activation. This systemic inflammatory response is composed of multiple components, and can be quantified by measuring markers of immune activation, inflammatory cytokines, acute phase reactants, endothelial activation markers, and markers of microbial translocation. This inflammation is clinically relevant, as it may contribute directly to HIV disease progression and non-AIDS related morbidity and mortality in HIV-infected patients. Because this inflammation persists even in the context of suppressive HAART, albeit at modestly decreased levels, adjunctive therapeutic strategies to attenuate this persistent inflammatory response are therefore needed. Herpes simplex virus type 2 is a common, clinically important co-infection seen in individuals living with HIV infection, and may contribute to this ongoing inflammation. This pilot trial will investigate whether short-term valacyclovir for HSV-2 suppression can decrease systemic inflammation in HAART-treated, HIV-1, HSV-2 co-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult (aged 18 years or older)
* documented HIV-1 infection (determined by EIA and Western blot)
* documented HSV-2 seropositivity (determined by ELISA during screening)
* no use of chronic anti-HSV therapy for the past 6 months, and not anticipated to require chronic anti-HSV therapy during the study
* sustained plasma HIV RNA<50 copies/mL on HAART for at least 12 months
* no active opportunistic infection for at least 12 months

Exclusion Criteria:

* hepatitis C co-infection
* hepatitis B co-infection
* pregnancy or actively planning to become pregnant
* receiving chemotherapy, chronic steroid therapy or other immunomodulatory medications (e.g. interferon, azathioprine, methotrexate, TNF-alpha antagonists, etc.)
* Estimated creatinine clearance <30 mL/min
* Other medical condition likely to cause death within 24 months
* Enrolled in any other interventional clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage activated CD8+ T-cells | 12 weeks
  Percentage of CD8+ T-cells co-expressing CD38 and HLA-DR

SECONDARY OUTCOMES:
Inflammatory markers | 12 weeks
  IL-6, hsCRP, sICAM-1, LPS
CD4 cell count | 12 weeks
  CD4 cell count (absolute and percentage)
Virologic blips | 12 weeks
  Plasma HIV RNA level >50 copies/mL but <1000 copies/mL, followed by a repeat plasma HIV RNA level <50 copies/mL.
Drug-related adverse events | 18 weeks
  Adverse events (AEs) are defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study medication. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not it is related to the medication.
HSV reactivations | 12 weeks
  Clinical reactivations of herpes simplex virus. Simultaneous reactivations at more than one anatomic site will be counted as a single reactivation event.
Acyclovir-resistant HSV | 18 weeks
  Clinical reactivations of herpes simplex virus that are microbiologically confirmed to be caused by acyclovir-resistant virus.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell HS Tan, MD FRCPC, Principal Investigator — University Health Network, University of Toronto; Sharon L Walmsley, MD FRCPC MSc, Principal Investigator — University Health Network, University of Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Result] Yi TJ, Walmsley S, Szadkowski L, Raboud J, Rajwans N, Shannon B, Kumar S, Kain KC, Kaul R, Tan DH. A randomized controlled pilot trial of valacyclovir for attenuating inflammation and immune activation in HIV/herpes simplex virus 2-coinfected adults on suppressive antiretroviral therapy. Clin Infect Dis. 2013 Nov;57(9):1331-8. doi: 10.1093/cid/cit539. Epub 2013 Aug 14. PMID 23946220
- See also: Study Results — http://www.ncbi.nlm.nih.gov/pubmed/23946220